CLINICAL TRIAL: NCT02908373
Title: Measuring Impact on Safety Culture in Nursing Homes, a Multifaceted Device for the Analysis of Care Associated Adverse Events
Brief Title: Risk Management in Nursing Homes
Acronym: EHPAGE
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC15_0053
Record Dates: First submitted 2016-09-12; First posted 2016-09-21 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Adverse Events Management in Nursing Homes
Keywords: risk management; nursing home; elderly; care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case group: Nursing homes benefiting first the implementation of the coaching model (methodological help for professionals on the patient safety culture): just after the first measure (overview of the situation)
  Interventions: Other: Implementation of the coaching model
- Control group: Nursing homes benefiting the implementation of the coaching model (methodological help for professionals on the patient safety culture): after the second measure (impact of the device on case group)
  Interventions: Other: Implementation of the coaching model

INTERVENTIONS:
Other: Implementation of the coaching model — 20 hours methodological help for each nursing home and an implementation kit

SUMMARY:
The Réseau QualiSanté (risk management network) hardly works on risk management in nursing homes. A model to help nursing homes managers to structure and analyze adverse events has been constructed by a working group of health professionals in the Réseau QualiSanté. Several questions appeared: is the model able to increase patient safety culture of professionals working in nursing homes? How to characterize adverse events in nursing homes? How frequent are they? The main objective of this research project EHPAGE is to measure the impact of the model to structure and analyze adverse events in nursing homes on the patient safety culture of professionals. The project combines quantitative data (questionnaire) and qualitative data (interviews).

DETAILED DESCRIPTION:
The main objective of this research project EHPAGE is to measure the impact of the model to structure and analyze adverse events in nursing homes on the patient safety culture of professionals. The coaching model is composed of a 20 hours methodological help for each nursing home and of an implementation kit.

To answer to the main objective, quantitative and qualitative data will be collected twice during the project: before the implementation of the coaching model and 12 months after.

Secondary objectives are:

1. To encourage the place of patient safety culture in strategic issues of nursing homes
2. To develop patient safety culture of professionals working in nursing homes
3. To develop a way to structure and make the reporting of adverse events in nursing homes more sustainable
4. To describe epidemiologic characteristic of adverse events in nursing homes
5. To propose a French validated questionnaire to evaluate patient safety culture reported by professionals in nursing homes An ancillary study is perform to describe epidemiologic characteristic of adverse events in nursing homes

ELIGIBILITY:
Inclusion Criteria:

* Nursing homes members of the Réseau QualiSanté (risk management network)
* Public or private legal status
* Agreeing to participate in the project

Exclusion Criteria:

* None

Ages: 65 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 61 nursing home located in Loire-Atlantique and Vendée departments in France. Loire-Atlantique and Vendée departments already benefit the risk management model from the réseau qualisanté located in Nantes University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1608 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

PRIMARY OUTCOMES:
impact of the coaching of the réseau QualiSanté: score expressed by the average percentages of positive responses to the "Overall perception of the safety of residents" dimension (= sum of 2 terms of positive response from the Likert scale) | 14 months after initial diagnosis.
  Initial analysis: estimate baseline characteristics of nursing homes (2 groups) Analysis of the primary endpoint primarily for professionals and secondly for nursing homes (consideration of cluster randomization)
  Professionals Analysis:
  Score of each professional "Overall perception of the safety of residents - OPOTSOR" dimension of NHSOPS questionnaire calculated for both measures in each arm Linear mixed model implemented to reflect the hierarchical data structure: score of the dimension "OPOTSOR" at assessment2 explained by the fixed effect group and the random effect of nursing homes.
  Adjustment with other variables if necessary Facility effect estimated with Intraclass correlation coefficient
  Nursing homes analysis:
  "Global perception of the safety of residents" dimension score of each nursing home calculated at assessment1 and 2 in each group Comparison of the average test scores at assessment2 for each nursing home

CONTACTS AND LOCATIONS:
Overall Officials: Leila MORET, MD PhD, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Teigne D, Mabileau G, Lucas M, Moret L, Terrien N. Safety culture in French nursing homes: A randomised controlled study to evaluate the effectiveness of a risk management intervention associated with care. PLoS One. 2022 Dec 1;17(12):e0277121. doi: 10.1371/journal.pone.0277121. eCollection 2022. PMID 36454806
- [Derived] Teigne D, Mabileau G, Anthoine E, Lucas M, Leclere B, Moret L, Terrien N. Transcultural adaptation and psychometric study of the French version of the nursing home survey on patient safety culture questionnaire. BMC Health Serv Res. 2019 Jul 15;19(1):490. doi: 10.1186/s12913-019-4333-5. PMID 31307443